CLINICAL TRIAL: NCT06130189
Title: The Impact of Nutrition, Physical Activity Habits and Adherence to the Mediterranean Diet on Children's Oral Health
Brief Title: Nutrition, Physical Activity, Mediterranean Diet Adherence, and Children's Oral Health
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, GÜLSEVİM ODA, Assistant professor, Ankara Medipol University
Other Study IDs: AnkaraMedipolGuls
Record Dates: First submitted 2023-11-07; First posted 2023-11-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Diet Habit; Family Characteristics; Tooth Decay; Periodontal Health
Keywords: children; dental caries; mediterranean diet; oral health
MeSH Terms: conditions — Feeding Behavior; Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main risk factors for dental caries are inadequate oral hygiene practices, cariogenic bacteria, and cariogenic diet. Among these factors, diet has a different dual relationship with dental caries. Dietary habits have the potential to be a risk factor for dental caries impaired oral and dental health can also lead to deficiencies in dietary intake.

Studies have shown that there is a decrease in gum and periodontal diseases in the adult age group with a diet compatible with the Mediterranean diet.

This cross-sectional study aims to examine the relationship between a diet compatible with the Mediterranean Diet and dental caries and gum health status in children. We hypothesize that children will have better gum health and less tooth decay with a diet compatible with the Mediterranean diet.

DETAILED DESCRIPTION:
Aim and Importance of the Research:

The Mediterranean diet (AD) is a healthy nutritional model, and the risk of major chronic inflammatory diseases decreases with a diet highly compatible with MD. It is thought that the protective effect of the Mediterranean diet is related to unsaturated fatty acids, the amount of dietary fiber, bioactive components, and antioxidants. It is known that diet affects the inflammatory reaction of periodontal tissues. It is stated that inflammatory reactions in the gums cannot develop, especially with a diet that does not contain refined carbohydrates. It is reported in the literature that reducing carbohydrate intake and taking additional Omega-3 fatty acids, vitamin C, vitamin D, antioxidants and fiber is beneficial for the health of periodontal tissues.

While excessive carbohydrate intake increases dysbiosis and chronic inflammatory diseases, a decrease in gingivitis has been observed by reducing carbohydrate intake. Dietary antioxidants play an important role in the development of adequate systemic reactions against oxidative stress. Clinical and in vitro studies have shown that antioxidants in the diet have positive effects on periodontal tissues.

Current studies report that there is a decrease in gum and periodontal diseases in the adult age group with a diet compatible with the Mediterranean diet. It is known that the Mediterranean diet reduces the amount of periodontopathogenic species, especially in supragingival plaque.

This cross-sectional study aims to examine the relationship between a diet compatible with the Mediterranean Diet and dental caries and gum health status in children. Secondly, the nutritional habits and behaviors of the family and the effects of the child's daily energy and nutrient intake on oral and dental health will be examined.

It is planned to include children between the ages of 0-14 who apply to Ankara Medipol University Oral and Dental Health Practice and Research Center Pedodontics Clinic. Parents of children who meet the study criteria will be informed about the research and an informed consent form will be obtained. Parents who volunteer to participate in the study will be asked to fill out the Demographic data form, Mediterranean Diet Quality Index (KIDMED), and Family Nutrition and Physical Activity (FNPA) screening tool. Additionally, a retrospective 24-hour food consumption record will be taken. Afterwards, oral and dental examinations of the children will be performed and the data obtained will be recorded.

Information on how to reach the participants: Families and children who meet the inclusion criteria and volunteer to participate in the study will be included in the patients who apply to the pedodontics clinic.

Forms used in data collection:

* Oral and dental examination indexes: Oral examinations of children will be performed by a single experienced pediatric dentist, using a mirror and probe, in the dentist's chair, and under appropriate lighting. Caries, extracted due to caries, filled primary and permanent teeth, and tooth surfaces in the child will be evaluated according to the caries index criteria of the World Health Organization (WHO-2013). Within the scope of evaluating plaque accumulation and gingival health, the plaque index (Silness & Löe, 1964) and gingival index (Löe & Silness, 1963) will be calculated.
* Mediterranean Diet Quality Scale (KIDMED):

Turkish validity and reliability study of the Mediterranean Diet Quality Scale in children was conducted by Şahingöz et al. (2019) . The scale consists of 16 questions, 12 of which have positive connotations and 4 of which have negative connotations. While positive answers to questions with negative connotations are scored as -1, positive answers to questions with positive connotations are scored as +1. As a result of the scoring, data ranging from 0-12 is obtained and evaluated in 3 main groups:

1. Those with ≥8 points optimal Mediterranean diet (good)
2. Scores between 4 and 7: Those whose compliance with the Mediterranean diet needs improvement (moderate)
3. If ≤3 points, very low nutritional quality (low)

   * Family Nutrition and Physical Activity screening tool (FNPA): The Family Nutrition and Physical Activity Screening Tool was developed by Ihmel et al. from Iowa State University in collaboration with the Academy of Nutrition and Dietetics (American Dietetic Association, ADA) in 2009. The original language of the FNPA scale is English. The FNPA scale is a behaviorally based assessment that evaluates family environments and combines information from a variety of behaviors associated with childhood obesity and was designed as a screening tool with potential for use by obesity researchers and a variety of clinical and public health professionals. The Turkish validity and reliability study was conducted by Ekici et al. (2021). The Turkish form of this tool consists of 20 items and is evaluated in a four-point Likert type. Each item is scored as 1 (never / rarely), 2 (sometimes), 3 (often) and 4 (very often / always). Six different items were reverse coded and these are items 3, 4, 5, 7, 10 and 13. The scores given to these items are summed up with the corresponding score in reverse order when calculating the total score (4; never / rarely, 3; sometimes, 2: often and 1; very often / always). The total score obtained from the scale varies between 20-80. Since there is no cut-off value when comparing the total score, high scores indicate less risky family practices and child behaviors for child obesity, while low scores indicate high-risk family environments and practices and child behaviors.
   * 24-hour retrospective food consumption record:The study will record individual daily food consumption with a "24-hour retrospective food consumption record" using the "Food Consumption Record Form".The researcher will ask the individuals included in the study about all the foods and drinks they consumed the day before, including their quantities. Daily energy and nutrient intakes of the individuals participating in the study will be calculated using the Nutrition Information Systems 8.2 program, and the percentages of daily energy intake, macro and micronutrients will be evaluated taking into account age and gender.

Sample size: The population of the study consists of healthy children between the ages of 0-14. The sample consists of healthy children who applied to Ankara Medipol University Oral and Dental Health Application and Research Center Pedodontics Clinic and those whose families volunteered to participate in the study. The sample size was calculated with G*Power 3.1.9.2. For this purpose, information obtained from previous similar studies (Sáenz-Ravello et al., 2023) was used as a reference. Considering the effect size as 0.25, the margin of error as 0.05, and the power value as 0.80, it was determined that at least 159 subjects were required.

Statistical Method(s):

The data obtained from the study will be evaluated with the SPSS 26.0 (Statistical Package for Social Science) statistical program. First of all, the distribution and skewness of the data will be evaluated with normality tests and will be expressed as mean (χ) and standard deviation (SD) or median (M), lower and upper values. Parametric (t-test) or non-parametric (Mann-Whitney U test) hypothesis tests are suitable for numerical/quantitative data when comparing the difference between two independent groups; For qualitative data, the appropriate chi-square test (Pearson/Fisher) will be used. Appropriate correlation analysis (Spearman/Pearson/Eta coefficient) will be performed to determine the relationship between numerical and qualitative variables. The value of p<0.05 will determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 3-14
* Not having a chronic/systemic disease (diabetes, allergies, etc.)
* Not having received radiotherapy or chemotherapy treatment
* Not having a mental or psychiatric disorder
* Agreeing to participate in the study

Exclusion Criteria:

* Over 14 years old and under 3 years old
* Having a chronic/systemic disease (diabetes, allergies, etc.)
* Having received radiotherapy or chemotherapy treatment
* Having a mental or psychiatric disorder
* Not agreeing to participate in the study

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: It is planned to include healthy children between the ages of 0-14 who apply to Ankara Medipol University Oral and Dental Health Practice and Research Center Pedodontics Clinic. Parents of children who meet the study criteria will be informed about the research and an informed consent form will be obtained.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Caries experiences | during enrollment once
  Oral examinations of children will be performed by a single experienced pediatric dentist, using a mirror and probe, in the dentist's chair, and under appropriate lighting. Caries, extracted due to caries, filled primary and permanent teeth, and tooth surfaces in the child will be evaluated according to the caries index criteria of the World Health Organization (WHO-2013).

SECONDARY OUTCOMES:
plaque index measurement | during enrollment once
  Oral examinations of children will be performed by a single experienced pediatric dentist, using a mirror and probe, in the dentist's chair, and under appropriate lighting. Within the scope of evaluating plaque accumulation the plaque index (Silness & Löe, 1964) will be calculated.
gingival index measurement | during enrollment once
  Oral examinations of children will be performed by a single experienced pediatric dentist, using a mirror and probe, in the dentist's chair, and under appropriate lighting. Within the scope of evaluating gingival health, the gingival index (Löe & Silness, 1963) will be calculated.
Mediterranean Diet Quality Scale (KIDMED): | during enrollment once
  The scale consists of 16 questions, 12 of which have positive connotations and 4 of which have negative connotations. While positive answers to questions with negative connotations are scored as -1 score, positive answers to questions with positive connotations are scored as +1 score. As a result of the scoring, data ranging from 0-12 is obtained and evaluated in 3 main groups: ≥8 points optimal Mediterranean diet (good), between 4 and 7: Those whose compliance with the Mediterranean diet needs improvement (moderate), ≤3 points, very low nutritional quality (low)b. Scores between 4 and 7: Those whose compliance with the Mediterranean diet needs improvement (moderate) c. If ≤3 points, very low nutritional quality (low)
  1. Those with ≥8 points optimal Mediterranean diet (good)
  2. Scores between 4 and 7: Those whose compliance with the Mediterranean diet needs improvement (moderate)
  3. If ≤3 points, very low nutritional quality (low)
Family Nutrition and Physical Activity screening tool (FNPA): | during enrollment once
  20 items :Each item is scored as 1 (never / rarely), 2 (sometimes), 3 (often) and 4 (very often / always). Six different items were reverse coded and these are items 3, 4, 5, 7, 10 and 13. The scores given to these items are summed up with the corresponding score in reverse order when calculating the total score (4; never / rarely, 3; sometimes, 2: often and 1; very often / always). The total score obtained from the scale varies between 20-80. Since there is no cut-off value when comparing the total score, high scores indicate less risky family practices and child behaviors for child obesity, while low scores indicate high-risk family environments and practices and child behaviors.
24-hour retrospective food consumption record: | during enrollment once
  The study will record individual daily food consumption with a "24-hour retrospective food consumption record" using the "Food Consumption Record Form".The researcher will ask the individuals included in the study about all the foods and drinks they consumed the day before, including their quantities. Daily energy and nutrient intakes of the individuals participating in the study will be calculated using the Nutrition Information Systems 8.2 program, and the percentages of daily energy intake, macro and micronutrients will be evaluated taking into account age and gender (16).

CONTACTS AND LOCATIONS:
Overall Officials: Gülsevim ODA, PhD, Principal Investigator — Ankara Medipol University Faculty of Dentistry; Merve Ekici, PhD, Principal Investigator — Department of Nutrition and Dietetics, University of Health Sciences
Locations (1):
- Ankara Medipol University Oral and Dental Health Practice and Research Center Pedodontics Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sofi F, Abbate R, Gensini GF, Casini A. Accruing evidence on benefits of adherence to the Mediterranean diet on health: an updated systematic review and meta-analysis. Am J Clin Nutr. 2010 Nov;92(5):1189-96. doi: 10.3945/ajcn.2010.29673. Epub 2010 Sep 1. PMID 20810976
- [Background] Bonaccio M, Di Castelnuovo A, Costanzo S, De Lucia F, Olivieri M, Donati MB, de Gaetano G, Iacoviello L, Bonanni A; Moli-sani Project Investigators. Nutrition knowledge is associated with higher adherence to Mediterranean diet and lower prevalence of obesity. Results from the Moli-sani study. Appetite. 2013 Sep;68:139-46. doi: 10.1016/j.appet.2013.04.026. Epub 2013 May 7. PMID 23665233
- [Background] Bosma-den Boer MM, van Wetten ML, Pruimboom L. Chronic inflammatory diseases are stimulated by current lifestyle: how diet, stress levels and medication prevent our body from recovering. Nutr Metab (Lond). 2012 Apr 17;9(1):32. doi: 10.1186/1743-7075-9-32. PMID 22510431
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Şahingöz, S. A., Özgen, L., & Yalçın, E. (2019). Akdeniz Diyet Kalitesi Ölçeğinin (Mediterranean Diet Quality-KIDMED) Geçerlik ve Güvenirlik Çalışması. Proceedings Book of 5th International Eurasian Congress on Natural Nutrition, Healthy Life & Sport, 1078-1088. 02-06 October 2019, Ankara/Turkey.
- [Background] Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM. Development and preliminary validation of a Family Nutrition and Physical Activity (FNPA) screening tool. Int J Behav Nutr Phys Act. 2009 Mar 12;6:14. doi: 10.1186/1479-5868-6-14. PMID 19284631
- [Background] Ekıcı, E. , Ikıısık, H. , Ankaralı, H. , Manav, G. , Colak, M. & Kozan, E. H. (2021). The validity and reliability of the Turkish version of the Family Nutrition and Physical Activity screening tool . Marmara Medical Journal , 34 (3) , 319-326 . DOI: 10.5472/marumj.1009125
- [Background] Pekcan, G. (2008). Beslenme durumunun saptanmasi. Diyet El Kitabi, 726, 67-141.
- [Result] Woelber JP, Bremer K, Vach K, Konig D, Hellwig E, Ratka-Kruger P, Al-Ahmad A, Tennert C. An oral health optimized diet can reduce gingival and periodontal inflammation in humans - a randomized controlled pilot study. BMC Oral Health. 2016 Jul 26;17(1):28. doi: 10.1186/s12903-016-0257-1. PMID 27460471
- [Result] Kim HS, Park JW, Yeo SI, Choi BJ, Suh JY. Effects of high glucose on cellular activity of periodontal ligament cells in vitro. Diabetes Res Clin Pract. 2006 Oct;74(1):41-7. doi: 10.1016/j.diabres.2006.03.034. Epub 2006 Jun 30. PMID 16814898
- [Result] Hujoel P. Dietary carbohydrates and dental-systemic diseases. J Dent Res. 2009 Jun;88(6):490-502. doi: 10.1177/0022034509337700. PMID 19587153
- [Result] Saenz-Ravello G, Matamala L, Cisternas P, Gamonal J, Hernandez P, Santos NCD, Deng K, Baeza M. Association between the Mediterranean Diet Index and self-reported Gingival Health Status Indicators in a population of Chilean adults: a cross-sectional study. J Appl Oral Sci. 2023 Jul 3;31:e20230100. doi: 10.1590/1678-7757-2023-0100. eCollection 2023. PMID 37403879
- [Result] Altun E, Walther C, Borof K, Petersen E, Lieske B, Kasapoudis D, Jalilvand N, Beikler T, Jagemann B, Zyriax BC, Aarabi G. Association between Dietary Pattern and Periodontitis-A Cross-Sectional Study. Nutrients. 2021 Nov 21;13(11):4167. doi: 10.3390/nu13114167. PMID 34836422
- [Result] Tennert C, Reinmuth AC, Bremer K, Al-Ahmad A, Karygianni L, Hellwig E, Vach K, Ratka-Kruger P, Wittmer A, Woelber JP. An oral health optimized diet reduces the load of potential cariogenic and periodontal bacterial species in the supragingival oral plaque: A randomized controlled pilot study. Microbiologyopen. 2020 Aug;9(8):e1056. doi: 10.1002/mbo3.1056. Epub 2020 May 17. PMID 32419378
- [Result] Laiola M, De Filippis F, Vitaglione P, Ercolini D. A Mediterranean Diet Intervention Reduces the Levels of Salivary Periodontopathogenic Bacteria in Overweight and Obese Subjects. Appl Environ Microbiol. 2020 Jun 2;86(12):e00777-20. doi: 10.1128/AEM.00777-20. Print 2020 Jun 2. PMID 32276980